CLINICAL TRIAL: NCT00321308
Title: A Randomized Phase II Trial Of Pemetrexed With Or Without PF-3512676 For The Treatment Of Patients With Locally Advanced Or Metastatic Non-Small Cell Lung Cancer After Failure Of One Prior Chemotherapy Regimen For Advanced Disease
Brief Title: Trial of Pemetrexed With or Without PF-3512676 in Advanced Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See Termination Reason in Detailed Description.
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A8501004
Record Dates: First submitted 2006-05-02; First posted 2006-05-03 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: advanced carcinoma, non-small cell lung cancer, phase II, pemetrexed, Alimta, PF-3512676, immunotherapy, immunomodulator
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed; ProMune

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- B (Active Comparator): Standard of care chemotherapy
  Interventions: Drug: pemetrexed
- A (Experimental): Standard of care chemotherapy plus experimental intervention (PF-3512676)
  Interventions: Drug: pemetrexed + PF-3512676

INTERVENTIONS:
Drug: pemetrexed — 500 mg/m2 intravenously Day 1 of each 21 day cycle until disease progression or unacceptable toxicity
  Other Names: Alimta
  Arms: B
Drug: pemetrexed + PF-3512676 — pemetrexed 500 mg/m2 intravenously Day 1 of each 21 day cycle until disease progression or unacceptable toxicity
  Other Names: Alimta
  Arms: A

SUMMARY:
To assess the efficacy and safety of PF-3512676 administered in combination with pemetrexed for the treatment of patients with locally advanced or metastatic NSCLC who have failed one prior chemotherapy regimen

DETAILED DESCRIPTION:
PF-3512676 dosing was stopped 21 June 2007 when Pfizer decided to stop the administration of PF-3512676 in all trials which combined PF-3512676 with cytotoxic chemotherapy. The decision was made subsequent to DSMC recommendation to close two phase III randomized trials in non-small cell lung cancer which also combined PF-3512676 with cytotoxic chemotherapy, citing lack of efficacy concerns as the primary reason with safety issues (sepsis, thrombocytopenia) also contributing to the decision. Subjects were allowed to complete standard of care treatment and protocol follow-up. Data collection was completed on 31 January 2008.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic NSCLC
* Measurable disease
* ECOG PS 0 or 1

Exclusion Criteria:

* Known CNS metastasis
* Pre-existing autoimmune or antibody mediated disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-09; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 110 Events

SECONDARY OUTCOMES:
Overall Survival | Time of death
Overall Safety Profile | 28 days post treatment
Patient Reported Outcome | End of Treatment
Time to Tumor Progression | End of treatment
Overall Objective Response Rate | Time of disease progressive disease
Duration of Response | Time of disease progression

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (18):
- United States (15):
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Bentonville, Arkansas
  - Pfizer Investigational Site, Fayetteville, Arkansas
  - Pfizer Investigational Site, Hudson, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Mahwah, New Jersey
  - Pfizer Investigational Site, Midland Park, New Jersey
  - Pfizer Investigational Site, Paramus, New Jersey
  - Pfizer Investigational Site, Westwood, New Jersey
  - Pfizer Investigational Site, Oneida, New York
  - Pfizer Investigational Site, Oswego, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Sylvania, Ohio
  - Pfizer Investigational Site, Seattle, Washington
- Germany (2):
  - Pfizer Investigational Site, Großhansdorf
  - Pfizer Investigational Site, Mannheim
- Pfizer Investigational Site, Torino, Italy

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8501004&StudyName=Trial%20of%20Pemetrexed%20With%20or%20Without%20PF-3512676%20in%20Advanced%20Non-Small%20Cell%20Lung%20Cancer